CLINICAL TRIAL: NCT02800070
Title: Clinical Pilot Study of Autologous Stem Cell Transplantation of Cluster of Differentiation 34 Positive (CD34+) Cells Engineered to Express Alpha-Galactosidase A in Patients With Fabry Disease
Brief Title: Autologous Stem Cell Transplantation of Cells Engineered to Express Alpha-Galactosidase A in Patients With Fabry Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-074
Record Dates: First submitted 2016-04-15; First posted 2016-06-15 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fabry Disease
Keywords: autologous stem cell transplant; gene therapy; Fabry disease; lentivirus; haematopoietic stem cell transplant
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients will receive Health Canada approved transduced autologous CD34+ cell product.
  Interventions: Biological: Lentivirus Alpha-gal A transduced stem cells

INTERVENTIONS:
Biological: Lentivirus Alpha-gal A transduced stem cells

SUMMARY:
This is a first-in-human study for the treatment of Fabry disease. Eligible patients will have an autologous stem cell transplantation using CD34+ cells that are transduced with the lentivirus vector containing the human alpha-gal A gene. The researchers of this study would like to see if the re-introduction of transduced cells will help increase the levels of alpha-gal A enzyme levels and to determine the safety and toxicity of autologous stem cell transplantation using CD34+ cells transduced with lentivirus vector containing the alpha-gal A gene. This study's objective is to determine the safety and toxicity of lentivirus alpha-gal A transduced CD34+ cells in adult males with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients 18-50 years of age at the time of enrollment
2. Diagnosis of Fabry disease (FD) as defined by very low or absent α-gal A activity
3. Classic FD Type I phenotype with alpha-galactosidase A (GLA) genotyping
4. Patients on enzyme replacement therapy (ERT) prior to enrollment
5. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
6. Adequate organ function within 21 days prior to Pre-Treatment Phase:
7. Willing and capable of signing and giving written informed consent in accordance with Research Ethics Board (REB) requirements
8. Willing to comply with all procedures outlined in the study protocol, cooperative with the protocol schedule, able to return for safety evaluation, or otherwise likely to complete the study
9. Willing to abstain from sexual activity or willing to use condoms during sexual intercourse from day of Melphalan administration on day -1 of Phase 3 until after 12 months follow-up post-transplant.
10. Willing to not donate sperm after receiving Melphalan. Sperm banking will be recommended to any patient who would like to father children in the future.

Exclusion Criteria:

1. Males with variant Fabry Disease.
2. Female gender
3. Use of immunosuppressive agents or any anticoagulant
4. Ongoing ERT-related infusion associated reactions of moderate-to-severe intensity
5. Presence of anti-agalsidase immunoglobulin (Ig)G antibodies above a threshold (5-fold above normal;) or evidence of high titre neutralizing antibodies
6. Blood test positive for Hepatitis B virus (HBV), Hepatitis C virus (HCV), human immunodeficiency virus (HIV), human T-cell lymphotropic virus type 1 (HTLV-1), human T-cell lymphotropic virus type 1 (HTLV-2), or Venereal Disease Research Laboratory test (VDRL; Transmissible Disease (TD) testing will be done in Pre-Treatment Phase 2 - see section 5.1 for full panel of TD tests. Patients will only be excluded from the study if positive for the TD tests listed here in this exclusion).
7. Uncontrolled bacterial, viral, or fungal infections
8. Prior malignancies except resected basal cell carcinoma
9. Chronic Kidney Disease (CKD) stage >2
10. History of heart failure or left ventricle ejection fraction (LVEF) <45% or moderate to severe diastolic dysfunction by standard criteria
11. Arrhythmia: bundle branch block, heart block degree II or III, atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, ventricular fibrillation, cardiac arrest, pacemaker, implantable cardiac defibrillator
12. Coronary artery disease with angina, prior myocardial infarction, percutaneous transluminal coronary angioplasty with or without stent, coronary artery bypass graft surgery, moderate to severe valvular heart disease, valve replacement surgery
13. Uncontrolled hypertension
14. Diabetes mellitus
15. Advanced liver disease, liver failure, cirrhosis
16. Immune deficiency state
17. Moderate-to-severe chronic obstructive pulmonary disease (COPD)
18. Any hematological condition with white blood cells (WBC) <3.0 x109/L, platelet count <100 x109/L, and/or hemoglobin <100 g/L
19. Prior bone marrow transplant (BMT) or organ transplant
20. Any condition that would preclude use of Melphalan
21. Use of a drug with cytotoxic or immunosuppressive effect within 60 days of trial entry
22. Uncontrolled psychiatric disorder
23. Active chronic infection
24. Prior tuberculosis
25. Any other serious concurrent disease
26. Cognitive impairment that would prevent informed consent
27. Use of an investigational drug within 30 days of stem cell transplant (SCT)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07; Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 years
  Safety measurement will be based on all clinical and laboratory assessment post-baseline. The assessment will be the frequency of clinically notable abnormal vital signs and laboratory values, and the frequency of treatment-related adverse events.

SECONDARY OUTCOMES:
Alpha-gal A enzyme activity levels | 5 years
  Increase in α-gal A enzyme activity within the plasma, leukocytes, and Bone marrow aspirate.
Gb3 levels | 5 years
  Reduction of Gb3 in plasma and urine
lyso-Gb3 levels | 5 years
  Reduction of lyso-Gb3 in plasma and urine
lyso-Gb3 analogue (-28) | 5 years
  Reduction of lyso-Gb3 (-28) in plasma and urine
lyso-Gb3 analogue (-2) | 5 years
  Reduction of lyso-Gb3 (-2) in plasma and urine
lyso-Gb3 analogue (+16) | 5 years
  Reduction of lyso-Gb3 (+16) in plasma and urine
lyso-Gb3 analogue (+34) | 5 years
  Reduction of lyso-Gb3 (+34) in plasma and urine
lyso-Gb3 analogue (+50) | 5 years
  Reduction of lyso-Gb3 (+50) in plasma and urine
vector copy number per genome on the CD34+ cell population | 5 years
  Persistence of LV-transduced cells as measured by quantitative (q)PCR
transduction efficiency | 5 years
  Vector copy number per genome on the CD34+ cell population
transduction efficiency | 5 years
  Number of colonies positive by PCR for the provirus out of number plated in the colony assay

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Alberta Children's Hospital, University of Calgary, Calgary, Alberta
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Khan A, Barber DL, Huang J, Rupar CA, Rip JW, Auray-Blais C, Boutin M, O'Hoski P, Gargulak K, McKillop WM, Fraser G, Wasim S, LeMoine K, Jelinski S, Chaudhry A, Prokopishyn N, Morel CF, Couban S, Duggan PR, Fowler DH, Keating A, West ML, Foley R, Medin JA. Lentivirus-mediated gene therapy for Fabry disease. Nat Commun. 2021 Feb 25;12(1):1178. doi: 10.1038/s41467-021-21371-5. PMID 33633114